CLINICAL TRIAL: NCT00686647
Title: AngioSculpt® Scoring Balloon Catheter Multi-Center Coronary Bifurcation Study
Brief Title: AngioSculpt® Coronary Bifurcation Study
Acronym: AGILITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AngioScore, Inc. (Industry)
Responsible Party: Gary Gershony, M.D., Chief Medical Officer, AngioScore, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASC-ST1210
Record Dates: First submitted 2008-05-28; First posted 2008-05-30 (Estimated); Results first posted 2011-08-10 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2011-07

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia
Keywords: Coronary Angioplasty; Coronary Stents; Scoring Balloons; Coronary Artery Bifurcation Lesions
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: AngioSculpt® Scoring Balloon Catheter — Use of a stent for the main branch of a bifurcation lesion and use of a scoring balloon for the side branch of the same bifurcation lesion
Device: AngioSculpt Scoring Balloon Catheter — Treatment of the side-branch vessel of true bifurcation lesions using the AngioSculpt device

SUMMARY:
The purpose of this study is to evaluate a new angioplasty catheter, AngioSculpt® for the treatment of bifurcation lesions (blockages occurring at branch points) in coronary arteries.

DETAILED DESCRIPTION:
Background: Bifurcation lesions, which consist of a narrowing occurring at branch points of coronary arteries, typically involve both the main branch (parent vessel) and an adjacent side branch. These lesions pose a particularly challenging situation for angioplasty procedures due to the difficulty of covering both branches with stents and a higher rate of recurrence (restenosis). A new angioplasty scoring balloon catheter (AngioSculpt®) has recently been approved for the treatment of narrowings in coronary arteries. The AngioSculpt® catheter incorporates a nitinol device that consists of spiral wires that wrap around the balloon catheter. As the balloon inflates, the spiral wires score the lesion allowing the balloon to be more stable (avoid slippage) and may enlarge the narrowed sections of the artery with less pressure or risk of dissection (uncontrolled tearing of the inner lining of the artery wall commonly seen with conventional balloons).

Study Purpose: To demonstrate the safety and efficacy of the AngioSculpt® used in conjunction with coronary stents (implantable wire mesh tubes for scaffolding blocked arteries) for the treatment of coronary artery bifurcation narrowings and to compare these results with the historical outcomes associated with the use of conventional balloons and stents in the treatment of bifurcation lesions.

Study Design: A prospective, multi-center, non-randomized, single-arm study with results compared to a literature search derived historical control for conventional balloon angioplasty (OPC - Objective Performance Criteria). The intent of this study is to enroll and treat 100 patients at 8 U.S. interventional cardiology programs with clinical follow-up planned at 30 days and 9 months following the procedure.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age and able to give informed consent.
* Patients with significant (> 50% diameter stenosis) native coronary artery disease involving a bifurcation and the ostium of the side branch vessel (Medina class (x, x, 1)) including stable or unstable angina and silent ischemia.
* Patients with lesions suitable for percutaneous coronary intervention (PCI).

Exclusion Criteria:

* Concomitant use of Rotablator, Cutting Balloon, or investigational coronary devices.
* Additional planned coronary interventions for a non-target lesion within 9 months of the study procedure.
* Left ventricular ejection fraction < 35%
* Patients refusing or not candidates for emergency coronary artery bypass grafting (CABG)surgery
* Uncontrolled severe hypertension (systolic BP >180 mm Hg or diastolic BP >110 mm Hg)
* Patients who are not candidates for chronic treatment with aspirin or Clopidogrel/Ticlopidine
* Severe renal failure with creatinine >2.0 mg/dL
* Untreated pre-procedural hemoglobin <10 g/dL
* Coagulopathy manifested by platelet count <100,000 or International Normalized ratio (INR) >2.0 (INR is only required in patients who have taken warfarin within 2 weeks of enrollment)
* Women who are known or suspected to be pregnant
* Patients in cardiogenic shock
* Acute myocardial infarction (MI) within the past 72 hours, and/or elevated CPK (and abnormal Troponin-I) at the time of enrollment
* Patients with a life expectancy of less than 1 year
* Target main branch vessel < 2.5 mm in diameter
* Target main branch lesion > 30 mm in length
* Intended use of a bare metal stent (BMS) in the main branch
* Target side branch vessel < 2.0 mm in diameter
* Target side branch lesion > 15 mm in length
* Target bifurcation angle > 90º (distal angle)
* Totally obstructed target coronary arteries (TIMI 0 or 1 flow)
* Target bifurcation lesion within a previously placed stent (i.e. in-stent restenosis (ISR))
* Target bifurcation lesion within a surgical conduit (e.g. saphenous vein or internal mammary)
* Target lesion demonstrating severe dissection prior to planned deployment of the AngioSculpt device
* Unprotected Left Main diameter stenosis ≥ 50%
* Visible thrombus (by angiography) at target lesion site
* Coronary spasm in the absence of a significant stenosis
* Patients who are concurrently participating in an investigational study when such participation could confound the treatment or outcomes of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2008-04; Primary Completion 2010-04 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey W. Moses, M.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Weisz G, Metzger DC, Liberman HA, O'Shaughnessy CD, Douglas JS Jr, Turco MA, Mehran R, Gershony G, Leon MB, Moses JW. A provisional strategy for treating true bifurcation lesions employing a scoring balloon for the side branch: final results of the AGILITY trial. Catheter Cardiovasc Interv. 2013 Sep 1;82(3):352-9. doi: 10.1002/ccd.24630. Epub 2013 Mar 9. PMID 22927100

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AngioSculpt Device
Started | 93
Completed | 91
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | AngioSculpt Device
Number analyzed (Participants) | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 57
  >=65 years | 36
Age Continuous [Mean (Standard Deviation); unit: years] | 61.54 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 67
Region of Enrollment [Number; unit: participants]
  United States | 93

OUTCOME MEASURES:

1. Primary Outcome: Procedural Success
Description: Defined as less than or equal to 30% diameter stenosis in the main branch and less than or equal to 70% diameter stenosis in the side branch at the conclusion of the procedure (including adjunctive stenting) in the absence of in-hospital major adverse cardiac events (MACE) [cardiac death, myocardial infarction (MI), or target lesion revascularization (TLR]
Time Frame: 1 day
Population: intention to treat
Measure: Number; unit: percentage of participants
Arm/Group | Overall Study
Number analyzed (Participants) | 93
percentage of participants | 91.4

2. Secondary Outcome: Major Adverse Cardiovascular Events
Description: cardiac death, myocardial infarction, or target lesion revascularization
Time Frame: 30 days
Population: intention to treat
Measure: Number; unit: percentage of particpants
Arm/Group | AngioSculpt Device
Number analyzed (Participants) | 93
percentage of particpants | 1.1

3. Secondary Outcome: Major Adverse Cardiac Events
Description: cardiac death, myocardial infarction, or target lesion revascularization
Time Frame: 9 months
Measure: Number; unit: percentage of participants
Arm/Group | AngioSculpt Device
Number analyzed (Participants) | 93
percentage of participants | 5.4

ADVERSE EVENTS:
Arm/Group | AngioSculpt Device
Serious Adverse Events (participants affected / at risk) | 2/93
Other Adverse Events (participants affected / at risk) | 7/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AngioSculpt Device (N=93)
cellulitis (Skin and subcutaneous tissue disorders) | 2 (2)
Death (Cardiac disorders) | 1 (1) — Investigator felt that patient death was due to arrythmia and not study related.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AngioSculpt Device (N=93)
Chest pain (Cardiac disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submission, the Sponsor, Institution, and Site Investigators will review and authorize the publication. A review period of 15 days for Presentational materials and abstracts; and 30 days for manuscripts is required for the Sponsor's review. Sponsor review does not include editorial privileges but can protect proprietary information and correct errors in data reporting or analysis if the Investigator agrees that there is an error.